CLINICAL TRIAL: NCT01969877
Title: A Randomized Multicenter Phase III Study of Cisplatin Plus Radiotherapy Compared to Cetuximab Plus Radiotherapy in Locally Advanced Head and Neck Cancer.
Brief Title: A Study of Cisplatin Plus Radiotherapy Compared to Cetuximab Plus Radiotherapy in Locally Advanced Head and Neck Cancer.
Acronym: ARTSCANIII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number 2012-001879-37; 2012-001879-37 (EudraCT Number)
Record Dates: First submitted 2013-10-16; First posted 2013-10-25 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Locally Advanced Head and Neck Cancer
Keywords: Head and neck cancer; Cetuximab; Cisplatin; Radiotherapy; Quality of life; Human papilloma virus; Health economy; Biomarker investigations
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental): Radiotherapy with a dose of 68.0 Gy in 34 fractions, and cetuximab with a loading dose of 400 mg/m2 one week before start of radiotherapy, then 250 mg/m2 weekly during radiotherapy (tumor stage 1-4).
  Interventions: Drug: cetuximab; Drug: cisplatin
- Arm 2 (Experimental): Radiotherapy with a dose of 73.1 Gy in 34 fractions, and cetuximab with a loading dose of 400 mg/m2 one week before start of radiotherapy, then 250 mg/m2 weekly during radiotherapy (tumor stage 3-4).
  Interventions: Drug: cetuximab; Drug: cisplatin
- Arm 3 (Experimental): Radiotherapy with a dose of 68.0 Gy in 34 fractions, and cisplatin weekly with a dose of 40 mg/m2 (tumor stage 1-4).
  Interventions: Drug: cetuximab; Drug: cisplatin
- Arm 4 (Experimental): Radiotherapy with a dose of 73.1 Gy in 34 fractions, and cisplatin weekly with a dose of 40 mg/m2 (tumor stage 3-4).
  Interventions: Drug: cetuximab; Drug: cisplatin

INTERVENTIONS:
Drug: cetuximab
Drug: cisplatin

SUMMARY:
The primary endpoint in this study is to investigate if there is a difference in overall survival in patients with locally advanced head and neck cancer, randomized to either radiotherapy and cetuximab or radiotherapy and cisplatin. A second randomization is performed in patients with T3-T4 tumors; allocated radiotherapy either 68.0 Gy or 73.1 Gy.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Histologically or cytologically confirmed , previous untreated head and neck squamous cell cancer of the oral cavity, hypopharynx, larynx or of the oral cavity aimed for unimodal treatment with radiotherapy with curative intent
* Tumor stage III and IV , but no evidence of distant metastases beyond the regional nodes in the neck
* WHO/Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* The patient must be expected to withstand radiotherapy combined with cisplatin or cetuximab
* The patient must be able to understand the information about the treatment and give a written informed concent to participate in the trial
* Adequate follow-up study must be possible; this will exclude a patient who is uncooperative
* Adequate renal function, creatinine clearance over 50 ml/min/1.73 estimated according to local practice at each study centre

Exclusion Criteria:

* Previous malignant disease in the head and neck region, with exception for basal cell carcinoma or curatively treated squamous cell carcinoma of the skin with follow-up time of at least 3 years
* Concomitant or previous malignancies. Exceptions are adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, or in situ carcinoma of the cervix uteri, or other previous malignancy with a disease-free interval of at least 5 years
* Two or more synchronous primary head and neck squamous cell cancer at time of diagnosis
* Co-existing disease prejudicing survival (expected survival less than 6 months)
* Absolute neutrophil count less than 1.5 x 109/L
* Platelet count less than 100 x 109/L
* Bilirubin over 1.5 times upper limit of normal
* Aspartate aminotransferase (ASAT) or Alanine aminotransferase (ALAT) more than 3 times upper limit of normal
* Pregnancy or lactation
* Allergy to study drug or to the excipients in their formulation
* Neuropathy grade 2 or more according to Common terminology criteria for adverse events (CTCAE) v.4.0
* Hearing loss/tinnitus is a relative exclusion criteria; the responsible physician decides whether the patient may be included in the study
* Severe cardiac illness; myocardial infarction within 6 months prior to randomization, severe congestive heart failure, severe cardiomyopathy, ventricular arrythmia, unstable angina, uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Overall survival | Every 3 month for 2 years, and every 6 month until 5 years for evaluation of overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gebre-Medhin, MD, PhD, Principal Investigator — Lund University Hospital
Locations (9):
- Sweden (9):
  - Gävle Hospital, Gävle
  - Sahlgrenska University Hospital, Gothenburg
  - County Hospital Ryhov, Jönköping
  - Central Hospital, Karlstad
  - University Hospital Linköping, Linköping
  - University Hospital Örebro, Örebro
  - Karolinska Universityhospital, Stockholm
  - Norrland University Hospital, Umeå
  - Västmanlands Hospital Västerås, Västerås

REFERENCES:
- [Derived] Gebre-Medhin M, Brun E, Engstrom P, Haugen Cange H, Hammarstedt-Nordenvall L, Reizenstein J, Nyman J, Abel E, Friesland S, Sjodin H, Carlsson H, Soderkvist K, Thomasson M, Zackrisson B, Nilsson P. ARTSCAN III: A Randomized Phase III Study Comparing Chemoradiotherapy With Cisplatin Versus Cetuximab in Patients With Locoregionally Advanced Head and Neck Squamous Cell Cancer. J Clin Oncol. 2021 Jan 1;39(1):38-47. doi: 10.1200/JCO.20.02072. Epub 2020 Oct 14. PMID 33052757